CLINICAL TRIAL: NCT04517968
Title: Evaluation of Immediate Implant Placement Using Customized Healing Abutment (Clinical Study)
Brief Title: Immediate Implant With Cusomized Healing Abutment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Immediate implants
Record Dates: First submitted 2020-08-14; First posted 2020-08-19 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Peri-implant Osteogensis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- immediate implant with customized healing abutment (Experimental)
  Interventions: Other: immediate implant with customized healing abutment

INTERVENTIONS:
Other: immediate implant with customized healing abutment — * All patients will be operated under local anesthesia.
  * Atraumatic extraction of the remaining root or tooth will be achieved.
  * A careful curettage of the socket will be performed if any granulation tissue is present.
  * Sequential drilling of the osteotomy site with copious irrigation will be done
  * The Implant is secured in place using a torque wrench.
  * Fabrication of the customized abutment with flowable composite by first placing a rubber dam between the abutment and the implant to prevent leakage of composite into the socket then start adding the composite in a manner to seal the socket.
  * Finishing the composite outside the patient's mouth will be done to ensure the borders are smooth with no sharp ends.
  * The abutment will be attached to the implant.

SUMMARY:
evaluate clinically and radiographically the effect of customized healing abutment on peri-implant osteogenesis following immediate implant placement.

DETAILED DESCRIPTION:
Now a day most people want to make immediate implant after extraction, which save them time and eliminates the need of second surgery. The problem is that the jummping gap between the implant and the bone that needs bone graft, this increase the cost on the patient. In this experiment we tend to evaluate this technique which may help us in growing autogenous bone and stop the need for bone grafting.

The aim of this study is to evaluate clinically and radiographically the effect of customized healing abutment on peri-implant osteogenesis following immediate implant placement.

A clinical trial was carried out on 8 patients (20-40 years old) with freshly extracted mandibular molars. Implants were placed immediately after extraction and a customized healing abutment will be fabricated. Patients were followed up clinically and radio graphically for 6 months.

ELIGIBILITY:
Inclusion criteria:

* Age range: 20 - 40 years
* Good oral hygiene
* A freshly extracted socket in the mandibular molar area.
* The gap between the implant and the bone will be at least 3-4 mm.

Exclusion criteria:

* Acute infection (periodontitis or mucosal infection)
* Patients on radiotherapy or chemotherapy.
* Alcohol or drug abuse.
* Patient with the systemic disorder (uncontrolled Diabetes mellitus, autoimmune diseases, bone diseases, etc.)
* Smokers.
* Parafunctional habits.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-02-03 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
change in bone density | at 3rd, 6th months
  Cone beam CT will be taken immediately and 6 months postoperatively On Demand 3d software** is used to assess:
  1. Crestal bone loss.
  2. Perapical Bone density.

SECONDARY OUTCOMES:
Change in pain | 1st day, 1 week, 4 weeks, 6 weeks, 12 weeks and after 6 months
  The patients will be examined using the Visual Analogue Scale (VAS). the scale is from 0-10 0 =no pain 10= most severe pain

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Alexandria, Egypt